CLINICAL TRIAL: NCT04101019
Title: Sphenopalatine Ganglion Block to Treat Shoulder Pain After Laparoscopic Surgery: A Prospective, Randomized, Double Blinded Trial
Brief Title: Sphenopalatine Ganglion Block to Treat Shoulder Pain After Laparoscopic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 421-19
Record Dates: First submitted 2019-07-08; First posted 2019-09-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-07

CONDITIONS: Nerve Block
MeSH Terms: interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Placebo Comparator): The patient will undergo the SPGB block with saline.
  Interventions: Drug: Saline Solution
- Active drug (Active Comparator): The patient will undergo the SPGB block with the active drug which will include 10% lidocaine diluted to 5%.
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Lidocaine — Intervention will include the SPGB block which will be performed by placing the patient supine with the neck extended and 1.5 ml of 5% lidocaine will be dripped into one or two nostrils.
  Arms: Active drug
Drug: Saline Solution — Intervention will include the SPGB block which will be performed by placing the patient supine with the neck extended and 1.5 ml of saline will be dripped into one or two nostrils.
  Arms: Control

SUMMARY:
This is a prospective double blinded randomized pilot trial to evaluate the efficacy of phenopalatine ganglion block (SPGB) block to manage shoulder tip pain (STP) after laparoscopic surgery.

Patients undergoing laparoscopic surgery will be approached by a member of the research team and those found eligible for participating will be enrolled after signing an informed consent form.

Patients will be randomized to have the SPGB block with saline versus active drug which contains 10% lidocaine diluted to 5%.

The block will be performed , by an experienced member of the research team, and the patient will then be followed up by the investigator for any adverse events and levels of shoulder pain.

DETAILED DESCRIPTION:
Purpose of the Study The purpose of this pilot study is to evaluate the efficacy of sphenopalatine ganglion block (SPGB) block to manage shoulder tip pain (STP) after laparoscopic surgery.

Background The laparoscopic technique has increasingly become a popular approach for many gynecologic, urologic, thoracic, bariatric and general surgical procedures. While laparoscopic surgery results in less postoperative pain than traditional open surgical techniques, it is associated with three distinct types of postoperative pain: incisional, visceral, and shoulder. The pain experienced in the shoulder is referred from irritation of the diaphragm and is referred to as shoulder tip pain (STP) to differentiate it from pain that originates in the shoulder. STP may persist for longer than incisional and visceral pain and may be the most difficult to treat. Narcotic and non-narcotic analgesics have only limited success in relieving STP, but none of these reliably eliminates STP, and they may be associated with undesirable systemic side effects. Recently the SPGB has been described as a means of managing STP (Grant 2018).

The SPGB was originally described more than 100 years ago as a treatment for headache (Sluder 1908). Since it was first described, the SPGB has been touted to relieve many types of pain, primarily of the head, but also pain extending down to the lower back (Berger 1986).

The SPG is located in pterygopalatine fossa adjacent to the sphenopalatine foramen. It is posterior to the middle nasal turbinate and separated from the nasal cavity by as little as 2 mm of mucosa. The proximity of the SPG to the nasal cavity facilitates renders it accessible to local anesthetic block. When local anesthetic is applied to the posterior nasopharyngeal mucosa, drug diffuses into the SPG and inhibits nerve conduction. The local anesthetic can be administered by injection, via a cotton-tipped applicator, or by simply dripping it into the nose when the patient is positioned with neck extension (Barre 1982).

Study Design This will be a randomized controlled trial to treat STP with local anesthetic or placebo in after laparoscopic surgery. The primary outcome variable will be reduction of STP.

Number of Subjects A power analysis was conducted to determine the minimum number of patents required to provide an indication that the SPG block will ameliorate STP after laparoscopic surgery. Assuming that a decrease in 2 NRS units will be clinically significant, and setting alpha as 0.05 and beta as 0.8, 36 patients per group will be needed, i.e., 76 total. The investigators will recruit 10% more patients to account for dropouts.

The investigators are therefore requesting approval to enroll 90 patients in the study.

(Tsai HW, Wang PH, Yen MS, Chao KC, Hsu TF, Chen YJ. Prevention of postlaparoscopic shoulder and upper abdominal pain: a randomized controlled trial. Obstet Gynecol. 2013 Mar;121(3):526-31).

Gender of Subjects This study is open to women and men.

Age of Subjects The study will be open to individuals aged 18 years old or greater.

Racial and Ethnic Origin There will be no effort to create a particular racial or ethnic distribution of patients for this study.

Inclusion Criteria

* Any type of gynecologic, urological, thoracic, bariatric and general surgical procedures
* Presence of post-operative STP, VAS > 4/10
* American Society of Anesthesiologists Class 1 - 3

Exclusion Criteria

* American Society of Anesthesiologists Class 4 or 5.
* Allergy to lidocaine.
* Any patient who the PI feels will be unable to comply with all protocol related procedures
* Shoulder pain prior to surgery

Methods & Procedures At any time during hospitalization after surgery (that is, once the patient is sufficiently awake to rate their pain in the ward until hospital discharge), if moderate-to-severe STP pain is present, the study team will be notified. The patient will be asked to rate their pain using an 11-point Numerical Rating Scale (NRS) to confirm that the VAS is > 4/10. Informed consent will then be obtained, and SPGB will be performed.

PROCEDURE:

Active drug and control:

Active drug group is 10% lidocaine diluted to 5% lidocaine (LIDO group). Control group is saline (SALINE group). The syringes will be filled (by the pharmacy?) with 1.5 mL of either solution and labeled in a blinded manner.

The SPGB will be performed by placing the patient supine with the neck extended, a position achieved by placing a padded support under their shoulders with the chip up. If the STP is unilateral, the head will be rotated to the side of the pain, and if the STP is bilateral, the head will be maintained in the midline position. Next, 1.5 mL of 5% lidocaine solution or saline will be dripped into one (for unilateral STP) or both nostrils (for bilateral STP), and the position will be maintained for 30 minutes. If the STP is not relieved, the procedure will be repeated using 1.5 mL of the active drug (5% lidocaine).

Patients will be followed after the SPG block(s), and the duration of pain relief will be monitored by serial assessments of the NRS. In addition, all patients will have PRN access to standard systemic analgesics as routinely ordered by their surgical service. Safety assessments will be performed on all subjects. Blood pressure, heart rate and respiratory rate will be obtained every 15 minutes after each SPG block for 90 minutes.

Data Analysis and Data Safety Monitoring Plan

The expected outcome of this study is a decrease in shoulder pain. A decrease in shoulder pain NRS of 2 points or greater will be taken as an indication that the block has worked.

Data collection

Additional data will be collected from an each of the study participant's electronic medical file. Data collection will include; demographic data, obstetric data, anesthetic data, anesthetic and surgical complications, analgesic requirements, hospital length of and admissions to ICU.

All gathered information will be coded in anonymous coding in order to preserve patient privacy rights.

Risk

The dripping of 5% lidocaine or saline into the nose is associated with minimal risk, but some discomfort.

The most common sources of discomfort are a sense of burning in the nasal mucosa when 5% lidocaine or saline is dripped into the nose. 5% lidocaine may produce a bitter taste in the mouth and numbness in the back of the throat as it drips down from the nasopharynx down into the oropharynx. Saline may produce a salty taste in the mouth as it drips down from the nasopharynx down into the oropharynx.

With any procedure that involves local anesthetic there is a risk of drug allergy, although this is a rare event.

Protection Against Risks To prevent and/or minimize potential risks or discomfort, the anesthesiologist who performs the SPGB will closely monitor the patient for the duration of administration of the block and for a minimum of 20 minutes following the block. Any annoying throat numbness or bitter taste would not be expected to last no more than 20 minutes or so after the last SPGB is performed. We are not aware of any risk to the patient from the intranasal administration of a maximum of 150 mg of lidocaine via the nose over 30 minutes. However, safety assessments will be performed on all subjects. Blood pressure, heart rate and respiratory rate will be obtained every 15 minutes after each SPG block for 90 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Any type of gynecologic, urologic, thoracic, bariatric and general surgical procedures
* Presence of post-operative STP, VAS > 4/10
* American Society of Anesthesiologists Class 1 - 3

Exclusion Criteria:

* American Society of Anesthesiologists Class 4 or 5.
* Allergy to lidocaine.
* Any patient who the PI feels will be unable to comply with all protocol related procedures
* Shoulder pain prior to surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
A numerical rate score decrease in shoulder pain | 90 minutes following performing the SPGB

CONTACTS AND LOCATIONS:
Locations (1):
- Beilinson hospital, Petach Tikvah, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Barre F. Cocaine as an abortive agent in cluster headache. Headache. 1982 Mar;22(2):69-73. doi: 10.1111/j.1526-4610.1982.hed2202069.x. No abstract available. PMID 7085264
- [Background] Berger JJ, Pyles ST, Saga-Rumley SA. Does topical anesthesia of the sphenopalatine ganglion with cocaine or lidocaine relieve low back pain? Anesth Analg. 1986 Jun;65(6):700-2. No abstract available. PMID 2871775
- [Background] Grant GJ, Echevarria GC, Lax J, Pass HI, Oshinsky ML. Sphenopalatine Ganglion Block to Treat Shoulder Tip Pain After Thoracic Surgery: Report of 2 Cases. A A Pract. 2018 Aug 15;11(4):90-92. doi: 10.1213/XAA.0000000000000746. PMID 29634542
- [Background] Tsai HW, Wang PH, Yen MS, Chao KC, Hsu TF, Chen YJ. Prevention of postlaparoscopic shoulder and upper abdominal pain: a randomized controlled trial. Obstet Gynecol. 2013 Mar;121(3):526-531. doi: 10.1097/AOG.0b013e318283fcca. PMID 23635614